CLINICAL TRIAL: NCT02124720
Title: Using Mobile Technology to Reduce Stereotypy in Children With Autism Spectrum Disorders
Brief Title: Using Mobile Technology to Reduce Stereotypy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Marc Lanovaz, Assistant Professor, Université de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERFAS-2014-15-030-P
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Child Development Disorders, Pervasive
Keywords: Autism spectrum disorders; Stereotypy; Repetitive behavior
MeSH Terms: conditions — Child Development Disorders, Pervasive; Autism Spectrum Disorder; Stereotypic Movement Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mobile application (Experimental): Use of the iSTIM mobile application 2 to 4 times per week over approximately 8 to 16 weeks
  Interventions: Behavioral: iSTIM

INTERVENTIONS:
Behavioral: iSTIM — Trained research assistants and parents will implement the assessments and interventions recommended by the iSTIM mobile application during sessions lasting between 10 and 60 minutes

SUMMARY:
Nearly all children with autism spectrum disorders engage in non-functional repetitive vocal and motor behaviours commonly referred to as stereotypy. These repetitive behaviours may considerably interfere with the child's daily functioning, learning, and social inclusion. As such, stereotypy generally has a negative impact on the child and family's health and quality of life. Several behavioural interventions have been developed to reduce engagement in stereotypy in children with autism spectrum disorders, but the limited number of specialists available, the long waiting lists associated with public health services in Canada, and the high costs of private services have considerably restricted accessibility. One potential solution to the limited availability and high costs of services is using a mobile application to recommend, teach, and monitor interventions designed to reduce engagement in stereotypy. To this end, the purpose of the study is to evaluate the effects of the iSTIM (i.e., individualized Stereotypy Treatment Integrated Modules), a mobile application designed to assist parents in reducing stereotypy in children with autism spectrum disorders. Specifically, we will assess whether the iSTIM correctly estimates the frequency or duration of stereotypy, offers suggestions consistent with recommended clinical practices, effectively reduces engagement in stereotypy, and is socially acceptable, safe, and easy to use for parents of children with autism spectrum disorders. The results of the study will allow us to determine whether the mobile application may be used to treat this core symptom in children with autism spectrum disorders, which could potentially reduce waiting times and costs of providing health services to this population. By reducing engagement in stereotypy, the iSTIM may also promote and facilitate the social participation as well as improve the quality of life and health of children with autism spectrum disorders and their families.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of autism spectrum disorders
* Must engage in at least one form of stereotypy

Exclusion Criteria:

* Stereotypy occurs less than 12 times per hour (or less than 20% of time)
* The form of stereotypy is potentially dangerous for the person (e.g., head banging, self-biting)
* The form of stereotypy is maintained by social consequences (e.g., attention, task avoidance)

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2014-12; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Frequency and duration of stereotypy | 2 to 4 times per week over 8 to 16 weeks
  Direct observation of the frequency and duration of stereotypy during 10- to 60-minute sessions

SECONDARY OUTCOMES:
Social validity score | Immediately following the end of the intervention (i.e., after 8 to 16 weeks)
  The user responds to a social validity questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Lanovaz, Ph.D., Principal Investigator — Université de Montréal
Locations (3):
- Canada (3):
  - Monarch House, Mississauga, Ontario
  - CRDITED de Montréal, Montreal, Quebec
  - Gold Centre, Montreal, Quebec